CLINICAL TRIAL: NCT01360957
Title: Effect of Consumption of Black Cumin (Nigella Sativa L.) Water Extract on Weight Loss in Overweight Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Mahnaz Kazemipoor has not handed over human subject review board approval letter to her colleague.
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Shahid Beheshti University of Medical Sciences, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23911
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2011-02

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Water flavored placebo (Placebo Comparator): to be given orally in a dosage of 30 ml trice daily for 60 days
  Interventions: Dietary Supplement: Black cumin water extract as a traditional medicine
- Black cumin water extract as a traditional medicine (Experimental): Black cumin water extract as a traditional medicine to be given orally in a dosage of 30 ml trice daily for 60 days
  Interventions: Dietary Supplement: Black cumin water extract as a traditional medicine

INTERVENTIONS:
Dietary Supplement: Black cumin water extract as a traditional medicine — to be given orally in a dosage of 30 ml trice daily for 60 days

SUMMARY:
The purpose of this clinical trial is to study the therapeutic effect of black cumin water extract (Nigella sativa L.) on obesity and overweight

DETAILED DESCRIPTION:
The worldwide prevalence of obesity has reached epidemic proportions mostly in low-income and transitional than in industrialized countries. Changes in dietary habits and sedentary lifestyles are known to be associated with changes in health and increased prevalence of chronic diseases in the population. The need to promote healthy nutrition for the population must be pursued vigorously, as the escalation of nutrition-related chronic degenerative diseases - once an urban phenomenon - has now spread to the rural population at an alarming rate. During the past decades efficacious strategies have been developed for prevention of these diseases. These strategies involve general lifestyle changes, which include, healthy diet, optimal weight, physical activity, moderate or no alcohol consumption, control of diabetes mellitus and in particular, treatment of obesity. Although the global market for satiety, fat burning and other weight management remedies has been grown, the awareness of the benefits of weight management ingredients is neither sufficient nor clearly perceived by consumer. Subsequently, the opportunities for scientifically-substantiated weight management ingredients regarding the natural and herbal dietary pattern are impressive.

The seed of Nigella sativa (black cumin) is one of the most common traditional herbs for weight loss in the Middle East which is usually used as a spice as well as traditional medicine to treat a variety of health conditions especially inflammatory diseases and obesity.

Furthermore, many of the components present in black cumin including polyphenols have been attributed to have anti-inflammatory and anti-obesity effect which further supports our hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Being Obese

Exclusion Criteria:

* Having heart disease or renal disease
* using drugs influencing metabolism and appetite

Ages: 16 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
BP (blood pressure) | 0 and12 weeks
  Change from Baseline in Systolic Blood Pressure at 12 weeks
HR (heart rate) | 0 and 12 weeks
  Change from Baseline in heart rate at 12 weeks
Body water (percentage) | 0 and 12 weeks
  Change from Baseline in body water at 12 weeks
Fat free mass (percentage) | 0 and 12 weeks
  Change from Baseline in fat free mass at 12 weeks
Fat mass (percentage) | 0 and 12 weeks
  Change from Baseline in fat mass at 12 weeks
Bone mass | 0 and 12 weeks
  Change from Baseline in bone mass at 12 weeks
BMR (basic metabolic rate) | 0 and12 weeks
  Change from Baseline in BMR at 12 weeks
AMR (active metabolic rate) | 0 and 12 weeks
  Change from Baseline in AMR at 12 weeks

SECONDARY OUTCOMES:
BMI (body mass index) | 0 and 12 weeks
  Change from Baseline in BMI at 12 weeks
WHR (waist to hip ratio) | 0 and 12 weeks
  Change from Baseline in WHR at 12 weeks
MUAC (mid upper arm circumference) | 0 and 12 weeks
  Change from Baseline in MUAC at 12 weeks
Wrist circumference | 0 and 12 weeks
  Change from Baseline in wrist circumference at 12 weeks
Changes in appetite as measured by a 10-point visual analog scale (VAS) | 0 and 12 weeks
  Change from Baseline in VAS at 12 weeks